CLINICAL TRIAL: NCT07197944
Title: A Phase 3, Double-blind, Randomized, Parallel Group, Placebo-controlled, Multicenter Trial to Confirm the Efficacy and Safety of Glepaglutide 10 mg Twice Weekly, Followed by a Long-term, Open-label Safety Evaluation in Patients With Short Bowel Syndrome-intestinal Failure (SBS-IF)
Brief Title: Efficacy And Safety Evaluation of Glepaglutide in Treatment of SBS
Acronym: EASE SBS 5
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zealand Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZP1848-23029; 2024-512486-14-00 (EU CTIS Number); U1111-1302-6092 (Other: UT Number)
Record Dates: First submitted 2025-09-26; First posted 2025-09-30 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Short Bowel Syndrome
Keywords: Intestinal Failure; Pathologic Processes; Malabsorption Syndromes; Intestinal Diseases; Gastrointestinal Diseases; Digestive System Diseases; Postoperative Complications; Short Bowel Syndrome; Syndrome
MeSH Terms: conditions — Short Bowel Syndrome; Intestinal Failure; Pathologic Processes; Malabsorption Syndromes; Intestinal Diseases; Gastrointestinal Diseases; Digestive System Diseases; Postoperative Complications; Syndrome

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two groups (arms) in parallel: one group receives glepaglutide, and the other group receives a placebo. After this initial phase, both groups receive open-label treatment with glepaglutide.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Glepaglutide Group (Experimental)
  Interventions: Drug: Glepaglutide
- Placebo Group (Placebo Comparator): Placebo for glepaglutide
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Glepaglutide — Subcutaneous (SC) injections twice weekly
  Other Names: ZP1848
  Arms: Glepaglutide Group
Other: Placebo — SC injections twice weekly
  Arms: Placebo Group

SUMMARY:
The purpose of the present Phase 3 trial is to confirm the efficacy and safety of glepaglutide 10 mg twice weekly in a patient population with SBS-IF and generate additional long-term safety data.

Glepaglutide is the International Nonproprietary Name and United States Adopted Name (USAN) for ZP1848.

DETAILED DESCRIPTION:
The trial is a phase 3, double-blind, randomized, parallel-group, placebo-controlled, multicenter trial to confirm the efficacy and safety of glepaglutide 10 mg twice weekly, followed by a long-term, open-label safety evaluation in patients with short bowel syndrome-intestinal failure (SBS-IF).

ELIGIBILITY:
Key Inclusion Criteria:

* Signed informed consent;
* Age of 18 to 90 years;
* A diagnosis of SBS, defined as having a small bowel with an estimated length of less than 200 cm (equal to 79 inches) in continuity (latest intestinal resection ≥6 months before screening);
* Stable PS need of ≥3 days per week;
* No restorative surgery planned during the trial period;
* Having a stoma or colon in continuity.

Key Exclusion Criteria:

* More than 2 SBS- or PS-related hospitalizations within 6 months before screening;
* Poorly controlled Inflammatory Bowel Disease (IBD) that is moderately or severely active or a fistula that can interfere with the measurements or examinations required in the trial;
* History of colorectal cancer or any other type of cancer (except for margin-free resected cutaneous basal, squamous cell carcinoma or adequately treated in situ cervical cancer) unless the patient has been disease-free for at least 5 years; ongoing bowel obstruction;
* BMI <18.5 kg/m^2.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-10-23 (Estimated); Study Completion 2032-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in weekly Parenteral Support (PS) volume | Baseline to Week 24

SECONDARY OUTCOMES:
Proportion of participants achieving clinical response | Baseline to Week 52
  Defined as achieving a reduction of at least 20% in weekly PS volume
Proportion of participants achieving clinical response | Baseline to Week 20 and Week 24
  Defined as achieving a reduction of at least 20% in weekly PS volume
Proportion of participants with a reduction in days on PS ≥1 day/week | Baseline to Week 52
Proportion of participants with a reduction in days on PS ≥1 day/week | Baseline to Week 24
Proportion of participants with a reduction of 100% weekly PS volume (weaned-off) | Baseline to Week 52
Proportion of participants with a reduction of 100% weekly PS volume (weaned-off) | Baseline to Week 24
Proportion of participants achieving 'much better' Patient Global Impression of Change (PGIC) status | Week 24
  PGIC scoring categories are: 'Much better', 'A little better', 'No change', 'A little worse', and 'Much worse'
Change in weekly PS volume | Baseline to Week 12
Change in weekly PS volume | Baseline to Week 8
Incidence of Treatment Emergent Adverse Events (TEAEs) | Baseline to Week 52

IPD SHARING:
Plan to Share IPD: No